CLINICAL TRIAL: NCT04584658
Title: Dysphagia and Dysphonia Outcomes in SARS CoV-2 (COVID-19): A Prospective Observational Cohort Study.
Brief Title: Dysphagia and Dysphonia Outcomes in SARS CoV-2 (COVID-19) Infection (DYADS Study)
Acronym: DYADS
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ekpemi Irune, Consultant Otolaryngology, Head & Neck Surgeon., Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 20/NW/0333
Record Dates: First submitted 2020-10-10; First posted 2020-10-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Dysphagia; Dysphonia; Subglottic Stenosis; Voice Disorders; Swallowing Disorder; Covid19; SARS (Severe Acute Respiratory Syndrome); SARS Pneumonia; Quality of Life; SARS-CoV-2 Infection
MeSH Terms: conditions — Deglutition Disorders; Dysphonia; Voice Disorders; COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fibreoptic Endoscopic Evaluation of Swallowing (FEES) — This is the use of endoscopy during feeding trials. The patient is fed different consistencies of food and drink while an endoscope is in place (usually passed through the nasal passage and down into the throat). The endoscope provides a bird's eye view to the transit of food through the upper aero-digestive tract. This provides information from the point of food bolus formation in the mouth to the movement of the base of the tongue; the movement of pharyngeal muscles; the deflection of the epiglottis to protect the airway including the closure of the vocal cords and the passage of food into the oesophagus. Any abnormality in these steps are noted during FEES. Liquids, thickened fluids, semi-solids and solids are some of the food textures that are tested.
Diagnostic Test: Videofluoroscopy — A radio opaque dye is used to label the test food and drink items offered to the patient. Following this, x-ray technology is used to create a video of the outline of the patient and the structures responsible for chewing and swallowing as they injest the test materials. The study is carried out in real time in the radiology department in conjunction with a radiographer and an SLT.
Other: Dysphagia Handicap Index (DHI) — This is a 25-item questionnaire assessing three domains: physical (9 items), functional (9 items), and emotional aspects (7 items) of the Quality of Life (QOL) in patients suffering with dysphagia. For each statement the patient checks if it applies to him/her all the time, some of the time or never. The suggested scores are 0, 2 and 4, respectively. Using this scoring system amounts to a DHI score range of 0 - 100. The higher the score, the worse the dysphagia related QOL. The patient is also asked to provide a rating of their own impression of the severity of the dysphagia experienced on a scale from 1 (normal) to 7 (severe problem).
Other: Voice Symptom Scale (VoiSS) — This is a 30-item validated quality of life tool that is also a self-reporting tool. It appraises the impact of the patient's abnormal voice from an emotional perspective, related physical symptoms and stratifies the impairment itself in context of day to day activities. VoiSS is currently the most psychometrically robust voice outcome measure. Each item is scored 0 - 4 on the frequency responses: never, occasionally, some of the time, most of the time, always. The total score of 120 measures general voice pathology which is made up of Impairment = maximum score of 60; Emotional = maximum score of 32; Physical = maximum score of 28.

SUMMARY:
This study examines the presence, severity and natural history of dysphagia and dysphonia in the post-extubation and severely unwell COVID-19 patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with a positive SARS CoV-2 test.
* Patients who have been diagnosed with dysphonia and/or dysphagia following COVID 19 treatment.
* Patients who require investigation and management for dysphonia and/or dysphagia following COVID 19 treatment.
* Adult patients aged 18 years - 85 years.
* Patients that meet threshold for referral to the joint MDT clinic following screening

Exclusion Criteria:

* Patients who cannot undertake the assessment for dysphonia and/or dysphagia.
* Patients who are being managed with palliative intent.
* Patients with pre-existing dysphonia and/or dysphagia not previously responding to therapy (pre-existing prior to COVID-19 diagnosis).

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients identified with dysphagia and dysphonia secondary to COVID19 infection. Specifically severely unwell patients and post-extubation patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is severity of dysphonia and dysphagia at the time of initial assessment t = day 0 (for ITU patients: Day 0 = 24 hours after extubation or decannulation). | t = day 0 (for ITU patients: Day 0 = 24 hours after extubation or decannulation).
  Based on therapy outcome measures from FEES, VoiS

SECONDARY OUTCOMES:
The severity of dysphonia and/or dysphagia over an initial 12 month period (at t = 14 days, 1 month, 3 months, 6 months, 9 months, 12 months) | t = 14 days, 1 month, 3 months, 6 months, 9 months, 12 months
  Clinical assessment including outcome measures, FEES and/or Videofluoroscopy
The severity of dysphonia and/or dysphagia at t = day 5, day 10, day 14, day 21 - For in-patients only. | t = day 5, day 10, day 14, day 21 - For in-patients only.
  Clinical assessment including outcome measures, FEES and/or Videofluoroscopy
Relationship between severity of dysphonia and/or dysphagia with grade of ARDS | t = day 0 and 9 months
  Clinical assessment including outcome measures, FEES and/or Videofluoroscopy
Relationship between severity of dysphonia and/or dysphagia with length of intubation | t = day 0 and 9 months
  Clinical assessment including outcome measures, FEES and/or Videofluoroscopy
Relationship between severity of dysphonia and/or dysphagia with duration of mechanical ventilation | t = day 0 and 9 months
  Clinical assessment including outcome measures, FEES and/or Videofluoroscopy
Relationship between severity of dysphonia on quality of life using Voice Symptom Scale (VoiSS) questionnaire over time at day 0, 1 month and 9 months. | t = day 0, 1 month and 9 months.
  Questionnaire assessment: This is a 30-item validated quality of life tool that is also a self-reporting tool. It appraises the impact of the patient's abnormal voice from an emotional perspective, related physical symptoms and stratifies the impairment itself in context of day to day activities. VoiSS is currently the most psychometrically robust voice outcome measure. Each item is scored 0 - 4 on the frequency responses: never, occasionally, some of the time, most of the time, always. The total score of 120 measures general voice pathology which is made up of Impairment = maximum score of 60; Emotional = maximum score of 32; Physical = maximum score of 28
Relationship between severity of dysphagia on quality of life using Dysphagia Handicap Index (DHI) questionnaire over time at day 0, 1 month and 9 months | t = day 0, 1 month and 9 months
  Questionnaire assessment: This is a 25-item questionnaire assessing three domains: physical (9 items), functional (9 items), and emotional aspects (7 items) of the Quality of Life (QOL) in patients suffering with dysphagia. For each statement the patient checks if it applies to him/her all the time, some of the time or never. The suggested scores are 0, 2 and 4, respectively. Using this scoring system amounts to a DHI score range of 0 - 100. The higher the score, the worse the dysphagia related QOL. The patient is also asked to provide a rating of their own impression of the severity of the dysphagia experienced on a scale from 1 (normal) to 7 (severe problem).

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No